CLINICAL TRIAL: NCT02797548
Title: Perioperative Antiplatelet Therapy in Patients With Drug-eluting Stent Undergoing Noncardiac Surgery
Acronym: ASSURE-DES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jung-min Ahn (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Jung-min Ahn, Assistant Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2016-10
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Antiplatelet Drugs
Keywords: drug-eluting stent; antiplatelet therapy; noncardiac surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin only (Experimental)
  Interventions: Drug: Aspirin only
- No antiplatelet therapy (Active Comparator)
  Interventions: Drug: No antiplatelet therapy

INTERVENTIONS:
Drug: Aspirin only — Aspirin only during surgery
  Arms: Aspirin only
Drug: No antiplatelet therapy — No antiplatelet therapy will be during surgery
  Arms: No antiplatelet therapy

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of perioperative antiplatelet therapy in patients with drug-eluting stent undergoing non-cardiac surgery.

DETAILED DESCRIPTION:
Subjects who can not be randomized due to any reason will be enrolled at observational group.

ELIGIBILITY:
Inclusion Criteria:

* Planned non-cardiac surgery at least after 12 months of implantation of drug eluting stent
* Low or intermediate risk level surgery
* Written informed consent

Exclusion Criteria:

* Acute coronary syndrome within 1 month
* Heart failure NYHA III to IV
* Contraindication to Aspirin
* On anticoagulant therapy
* Emergent surgery
* Cardiac surgery
* High bleeding risk surgeries, e.g., Intra-cranial surgery, Intra-spinal surgery, Retinal surgery
* Pregnancy or breast-feeding
* Life expectancy less than 1year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
The event rate of composite event of all-cause death, stent thrombosis, myocardial infarction, and stroke | 30 days
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event that is considered to have occurred if any one of several different events is observed.

SECONDARY OUTCOMES:
The event rate of all cause death | 30 days
The event rate of cardiac death | 30 days
The event rate of myocardial infarction | 30 days
The event rate of stroke | 30 days
The event rate of stent thrombosis | 30 days
The event rate of repeat revascularization | 30 days
The event rate of life threatening bleeding | 30 days
The event rate of major bleeding | 30 days
Quality of life score assessed by the EQ-5D-5L | 30 days
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  Higher score of EQ-5D and EQ VAS means the low quality of life. EQ-5D: the minimum and maximum values are 5 and 25 respectively. EQ VAS: the minimum and maximum values are 0 and 100 respectively.
Quality of life score assessed by Health-related Quality of Life Instrument with 8 Items (HINT-8) | 30 days
  HINT-8 was developed based on 4 health dimensions: physical, mental, social, and positive health dimensions. It consists of climbing stairs, endurance to pain, vitality, working, depression, memory, sleep, and happiness.
  Higher score of HINT-8 means the high quality of life. The minimum and maximum values are 0 and 100 respectively if convert to a percentage.
Cost-effective analysis | 30 days
  Cost-effective analysis based on average treatment costs for two perioperative antiplatelet therapy_Aspirin only vs. No antiplatelet therapy_in patients with drug-eluting stent undergoing non-cardiac surgery.

CONTACTS AND LOCATIONS:
Locations (35):
- Jaslok Hospital, Mumbai, India
- South Korea (32):
  - Asan Medical Center, Seoul, Songpa-gu
  - Hallym University Sacred Heart Hospital, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Dong-A Medical Center, Busan
  - Pusan National University Yangsan Hospital, Busan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Chungbuk National University Hospital, Cheonju
  - Gangwon National Univ. Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon St. Mary's Hosptial, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Wonkwang University Sanbon Hospital, Gunpo
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Wonkwang University Hospital, Iksan
  - National Health Insurance Service Ilsan Hospital, Ilsan
  - Pusan National University Hospital, Pusan
  - Sejong Chungnam National University Hospital, Sejong
  - Ewha Womans University Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
  - Yongin Severance Hospital, Yŏngin
- Turkey (Türkiye) (2):
  - Bagcilar Education and Training Hospital, Istanbul
  - SBU Bakirkoy Dr.Sadi Konuk Education and Training Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang DY, Lee SH, Lee SW, Lee CH, Kim C, Jang JY, Mehta N, Oh JH, Cho YR, Yoon KH, Ahn SG, Lee JH, Cho DK, Kim Y, Kim J, Cho GH, Lee KS, Park H, Vural M, Lim YH, Park KH, Lee BK, Lee JY, Park HW, Yoon YH, Lee JH, Lee SY, Park KW, Kang J, Kim HK, Kang SH, Park JH, Choi IC, Yu CS, Yun SC, Park DW, Hong MK, Park SJ, Kim JS, Ahn JM; ASSURE DES Investigators. Aspirin Monotherapy vs No Antiplatelet Therapy in Stable Patients With Coronary Stents Undergoing Low-to-Intermediate Risk Noncardiac Surgery. J Am Coll Cardiol. 2024 Dec 10;84(24):2380-2389. doi: 10.1016/j.jacc.2024.08.024. Epub 2024 Aug 31. PMID 39217573